CLINICAL TRIAL: NCT02914769
Title: Antidepressant Effects of Ayahuasca: a Randomized Placebo Controlled Trial in Treatment Resistant Depression
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Universidade Federal do Rio Grande do Norte (Other)
Collaborators: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, Draulio Barros de Araujo, Professor, Universidade Federal do Rio Grande do Norte
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CNPq-466760/2014-0
Record Dates: First submitted 2016-09-21; First posted 2016-09-26 (Estimated); Results first posted 2025-04-06 (Actual); Last update posted 2025-04-06 (Actual); Status verified 2025-04

CONDITIONS: Major Depression
Keywords: Depression; Ayahuasca; Psychedelics
MeSH Terms: conditions — Depressive Disorder, Major; Depression | interventions — Therapeutics

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- placebo (Placebo Comparator): patients receiving a passive placebo
  Interventions: Drug: placebo
- Ayahuasca (Experimental): patients receiving Ayahuasca
  Interventions: Drug: Ayahuasca

INTERVENTIONS:
Drug: Ayahuasca — patients will receive a single dose of ayahuasca.
  Other Names: treatment
  Arms: Ayahuasca
Drug: placebo — patients will receive a single dose of a passive placebo.
  Arms: placebo

SUMMARY:
The purpose of the present trial is to test the efficacy of Ayahuasca in treatment-resistant depression. Ayahuasca is a decoction of two plants, long used by Amazonian Amerindians. Traditionally, it is prepared by decoction of a bush (Psychotria viridis) with a liana (Banisteriopsis caapi). P. viridis is a rich source of N,N-dimethyltryptamine (DMT), a serotonergic agonist, and B. caapi contains potent monoamine oxidase-A inhibitors (MAOi-A), such as harmine, harmaline. The study is designed as a randomized placebo controlled trial with two parallel arms, and it will also evaluate changes of different biomarkers of depression including anatomical and functional Magnetic Resonance Imaging (MRI), serum levels of BDNF, TNF-a, cortisol, IL-6, and IL-10, polysomnography, neuropsychological, psychiatric scales and questionnaires.

DETAILED DESCRIPTION:
1) Background

The therapeutic effectiveness of currently available antidepressant is low. Less than 50% of the patients achieve remission after single treatment, and about 30% after four different treatments. Besides low response rates, pharmacological treatment are associated with several side effects and response onset is usually long (~2-3 weeks). Thus, great effort has been made to the development of alternative antidepressants. For instance, ketamine, a N-methyl-D-aspartate (NMDA) receptor antagonist, has rapid and potent antidepressant effects in treatment of major depressive and bipolar disorders.

This proposal aims at testing the antidepressant effects of Ayahuasca, traditionally prepared by decoction of two plants: Psychotria viridis and Banisteriopsis caapi, long used by Amazonian Amerindians. P. viridis is a rich source of the serotonergic agonist N,N-dimethyltryptamine (DMT), whereas B. caapi contains potent monoamine oxidase-A inhibitors (MAOi-A) such as harmine, harmaline, and tetrahydroharmine, a serotonin reuptake inhibitor.

Common effects of Ayahuasca include sedation, gastrointestinal distress, changes of spatiotemporal scaling, dissociation, sense of well-being, insights, feelings of apprehension, increased interoceptive attention and sensory pseudo-hallucinations. Effects begin at 30-40 min after oral intake, and last up to 4 hours. Previous studies suggest the absence of psychological, neuropsychological or psychiatric harm caused by prolonged Ayahuasca consumption, and it is not addictive, on the contrary, it also shows promise in treating addiction.

Recently, two preliminary open label studies have tested tolerability, safety and the antidepressant effect of Ayahuasca in treatment-resistant depression. In the first study, six patients were recruited, in the second, 17 patients. The results show significant decrease in depression severity (HAM-D & MADRS scales) already at 2 hours after intake, which lasted for 21 days. Although the results are promising, they must be considered with caution, specially due to the lack of control of the placebo effect, which is generally high in clinical trials.

Thus, the present study is a randomized placebo-controlled trial in 50 patients with treatment resistant depression. Besides the Antidepressant effects of Ayahuasca, this study will also evaluate different biomarkers of depression, including anatomical and functional Magnetic Resonance Imaging (MRI), serum levels of BDNF, TNF-a, cortisol, IL-6, and IL-10, polysomnography, neuropsychological and psychiatric scales and questionnaires.

2. Methods

All 50 patients will undergo routine evaluation, including complete blood testing for individual glycemic profile, serum cholesterol and triglyceride, plasma sodium and potassium, urea and creatinine.

Patients will undergo a wash-out period, between 7 and 14 days prior to the experimental session, depending on the lifetime of the antidepressant in use. Experiments will take place at the Hospital Universitário Onofre Lopes, a tertiary university hospital affiliated to the Universidade Federal do Rio Grande do Norte (UFRN), Brazil.

In the treatment session, 25 patients will drink Ayahuasca, 25 will drink an inert placebo. Psychiatric scales (HAM-D, MADRS, BPRS, CADSS and YMRS) will be completed during treatment session, day one before (-D1), one day after (+D1), two days (+D2), seven days (+D7), fourteen days (+D14), one month (+M1), and up to six months (+M6) following the treatment session. The following exams will also be conducted at D-1 and D+1: neuropsychological tests (watch test, trail test, and N-back), structural and functional MRI, polysomnography and blood testing (BDNF, TNF-a, cortisol, oxytocin, IL-6, and IL-10).

ELIGIBILITY:
Inclusion Criteria:

* Age: 18-60 years old;
* Diagnostic of major depressive disorder (DSM-IV);
* At least two previous unsuccessful antidepressant medications;
* Current depressive episode (HAM-D >= 17).

Exclusion Criteria:

* History of psychosis;
* Present or past history of bipolar disorder or schizophrenia;
* Diagnosis of current clinical disease, based on history, physical examination and routine hematologic and biochemical tests;
* Serious and imminent suicidal risk;
* Pregnancy, current drug or alcohol dependence;
* Previous experience with ayahuasca.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 35 (Actual)
Dates: Start 2014-02; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Draulio B de Araujo, Ph.D, Principal Investigator — Brain Institute - UFRN
Locations (1):
- Draulio B de Araujo, Natal, Rio Grande do Norte, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sanches RF, de Lima Osorio F, Dos Santos RG, Macedo LR, Maia-de-Oliveira JP, Wichert-Ana L, de Araujo DB, Riba J, Crippa JA, Hallak JE. Antidepressant Effects of a Single Dose of Ayahuasca in Patients With Recurrent Depression: A SPECT Study. J Clin Psychopharmacol. 2016 Feb;36(1):77-81. doi: 10.1097/JCP.0000000000000436. PMID 26650973
- [Background] Osorio Fde L, Sanches RF, Macedo LR, Santos RG, Maia-de-Oliveira JP, Wichert-Ana L, Araujo DB, Riba J, Crippa JA, Hallak JE. Antidepressant effects of a single dose of ayahuasca in patients with recurrent depression: a preliminary report. Braz J Psychiatry. 2015 Jan-Mar;37(1):13-20. doi: 10.1590/1516-4446-2014-1496. PMID 25806551
- [Derived] Zeifman RJ, Palhano-Fontes F, Hallak J, Arcoverde E, Maia-Oliveira JP, Araujo DB. The Impact of Ayahuasca on Suicidality: Results From a Randomized Controlled Trial. Front Pharmacol. 2019 Nov 19;10:1325. doi: 10.3389/fphar.2019.01325. eCollection 2019. PMID 31798447
- [Derived] de Almeida RN, Galvao ACM, da Silva FS, Silva EADS, Palhano-Fontes F, Maia-de-Oliveira JP, de Araujo LB, Lobao-Soares B, Galvao-Coelho NL. Modulation of Serum Brain-Derived Neurotrophic Factor by a Single Dose of Ayahuasca: Observation From a Randomized Controlled Trial. Front Psychol. 2019 Jun 4;10:1234. doi: 10.3389/fpsyg.2019.01234. eCollection 2019. PMID 31231276
- [Derived] Palhano-Fontes F, Barreto D, Onias H, Andrade KC, Novaes MM, Pessoa JA, Mota-Rolim SA, Osorio FL, Sanches R, Dos Santos RG, Tofoli LF, de Oliveira Silveira G, Yonamine M, Riba J, Santos FR, Silva-Junior AA, Alchieri JC, Galvao-Coelho NL, Lobao-Soares B, Hallak JEC, Arcoverde E, Maia-de-Oliveira JP, Araujo DB. Rapid antidepressant effects of the psychedelic ayahuasca in treatment-resistant depression: a randomized placebo-controlled trial. Psychol Med. 2019 Mar;49(4):655-663. doi: 10.1017/S0033291718001356. Epub 2018 Jun 15. PMID 29903051

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were recruited from psychiatrist referrals at local outpatient psychiatric units or through media advertisements. All procedures took place at the Onofre Lopes University Hospital (HUOL), Natal-RN, Brazil.
Pre-assignment Details: From January 2014 to June 2016, we assessed 218 patients for eligibility, and 35 met criteria for the trial. 183 patients not met inclusion criteria for the trial, 26 declined to participate and 14 were not enrolled due to other reasons (several clinical conditions).
Groups:
- Placebo: patients receiving a passive placebo
  placebo: patients will receive a single dose of a placebo.
Period: Overall Study
Arm/Group | Placebo | Ayahuasca
Started | 18 | 17
Completed | 15 | 14
Not Completed | 3 | 3
Not completed — Protocol Violation | 3 | 2
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Population: 218 patients were assessed for eligibility, and 35 met criteria for the trial. Six subjects had to be excluded: five no longer met criteria for depression in the day of dosing, and one dropped out before dosing.
Groups:
- Placebo: placebo: patients will receive a single dose of a placebo.
- Total: Total of all reporting groups
Arm/Group | Placebo | Ayahuasca | Total
Number analyzed (Participants) | 15 | 14 | 29
Age, Continuous [Mean (Standard Deviation); unit: years] | 39.71 (11.26) | 44.20 (11.98) | 41.95 (11.62)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 11 | 21
  Male | 5 | 3 | 8
Region of Enrollment [Count of Participants; unit: Participants]
  Brazil | 15 | 14 | 29
MADRS [Mean (Standard Deviation); unit: score] — This scale measures depression severity. Each item yields a score of 0 to 6; the overall score thus ranges from 0 to 60. Higher MADRS score indicates more severe depression.
  Usual cutoff points are a total score ranging from: 0 to 6 indicates that the patient is in the normal range (no depression); 7 to 19 indicates "mild depression"; 20 to 34 indicates "moderate depression"; a score of 35 and greater indicates "severe depression".
  score | 30.13 (5.55) | 36.14 (6.12) | 33.13 (5.83)
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 15 | 14 | 29
  Not Hispanic or Latino | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Hamilton Depression Rating Scale (HAM-D) Effect Seven Days After Dosing (D7)
Description: changes in depression severity, assessed by the Hamilton Depression Rating Scale (HAM-D) scale, from baseline to 7 days after dosing.
  Minimum and maximum scores are 0 and 50, respectively. Although the HAM-D form lists 21 items, the scoring is based on the first 17. Eight items are scored on a 5-point scale, ranging from 0 = not present to 4 = severe. Nine items are scored from 0-2.
  Lower HAM-D score indicates less severe depression (better outcome). Usual cutoff points are a total score ranging from: 0 to 7 indicates that the patient is in the normal range (no depression); 8 to 16 indicates "mild depression"; 17 to 23 indicates "moderate depression"; a score of 24 and greater indicates "severe depression".
Time Frame: seven days after dosing
Population: A fixed-effects linear mixed model, with baseline scores as covariate, examined changes in HAM-D at D7. Herein we report mean HAM-D scores at D7.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo | Ayahuasca
Number analyzed (Participants) | 15 | 14
score on a scale | 16.92 (7.36) | 9.72 (7.39)

2. Secondary Outcome: Montgomery-Asberg Depression Rating Scale (MADRS) Effect at D1, D2 and D7
Description: changes in depression severity, assessed by Montgomery-Asberg Depression Rating Scale (MADRS scale), from baseline to 1 day, 2 days, and 7 days after dosing. Lower MADRS score indicates less severe depression (better outcome).
  Minimum and maximum scores are 0 and 60, respectively. Usual cutoff points are a total score ranging from: 0 to 6 indicates that the patient is in the normal range (no depression); 7 to 19 indicates "mild depression"; 20 to 34 indicates "moderate depression"; a score of 35 and greater indicates "severe depression".
Time Frame: one, two and seven days after dosing
Population: Herein we report MADRS scores at D1, D2 and D7.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo | Ayahuasca
Number analyzed (Participants) | 15 | 14
score on a scale
  MADRS Scores at D1 | 21.49 (10.90) | 12.65 (10.27)
  MADRS Scores at D2 | 19.09 (10.44) | 10.32 (10.44)
  MADRS Scores at D7 | 26.76 (10.11) | 11.58 (10.27)

3. Secondary Outcome: Number of Participants With Reduction of 50% or More in Hamilton Depression Rating Scale(HAM-D) Scores at D7
Description: Response Rate:Number of Participants with reduction of 50% or more in Hamilton Depression Rating Scale (HAM-D) in baseline scores, assessed seven days after dosing.
Time Frame: seven days after dosing
Population: Response rate
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Ayahuasca
Number analyzed (Participants) | 15 | 14
Participants | 3 | 8

4. Secondary Outcome: Number of Participants With Reduction of 50% or More in Montgomery-Asberg Depression Rating Scale (MADRS) at D1, D2 and D7
Description: response rate: reduction of 50% or more in baseline scores, assessed at one day, two days and seven days after dosing by the MADRS scale.
Time Frame: one, two, and seven days after dosing
Population: Response rate
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Ayahuasca
Number analyzed (Participants) | 15 | 14
Participants
  D1 | 7 | 7
  D2 | 10 | 11
  D7 | 4 | 9

5. Secondary Outcome: Number of Participants With a Score Lower Then or Equal to 7 in the Hamilton Depression Rating Scale (HAM-D) at D7
Description: Number of Participants With a score lower then or equal to 7 in the Hamilton Depression Rating Scale (HAM-D) at seven days after dosing.
Time Frame: seven days after dosing
Population: Remission rate
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Ayahuasca
Number analyzed (Participants) | 15 | 14
Participants | 2 | 6

6. Secondary Outcome: Number of Participants With a Score Lower Then or Equal to 10 in the Montgomery-Asberg Depression Rating Scale (MADRS) at D1, D2 and D7
Description: Number of Participants With a Score Lower Then or Equal to 10 in the Montgomery-Asberg Depression Rating Scale (MADRS) at one, two and seven days after dosing.
Time Frame: one, two and seven days after dosing
Population: Remission rate
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Ayahuasca
Number analyzed (Participants) | 15 | 14
Participants
  D1 | 7 | 6
  D2 | 8 | 4
  D7 | 1 | 5

ADVERSE EVENTS:
Time Frame: One week.
Description: Definitions do not differ from the clinicaltrials.gov
Arm/Group | Placebo | Ayahuasca
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/14
Other Adverse Events (participants affected / at risk) | 4/15 | 10/14
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=15) | Ayahuasca (N=14)
Nausea (Gastrointestinal disorders) | 4 | 10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes